CLINICAL TRIAL: NCT07133035
Title: Investigation of Respiratory Function, Biomechanical Properties of Neck and Jaw Muscles and Pain Sensitivity in Individuals With Bruxism
Brief Title: Investigation of Respiratory Function in Bruxism
Status: Active, not recruiting | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, Seval Yilmaz, Principal Investigator, Atılım University
Other Study IDs: 6040102284-Bruxism
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Bruxism; Sleep
Keywords: bruxism; sleep; respiratory function; headache
MeSH Terms: conditions — Bruxism; Respiratory Aspiration; Headache | interventions — Respiratory Function Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bruxism: Individuals diagnosed with bruxism
  Interventions: Diagnostic Test: Pulmonary function test; Diagnostic Test: Fonseca Anamnestic Index; Other: Jenkins Sleep Scale; Other: Berlin Questionnaire; Other: Headache Impact Test-6
- Control: healthy individuals
  Interventions: Diagnostic Test: Pulmonary function test; Diagnostic Test: Fonseca Anamnestic Index; Other: Jenkins Sleep Scale; Other: Berlin Questionnaire; Other: Headache Impact Test-6

INTERVENTIONS:
Diagnostic Test: Pulmonary function test — Participants' respiratory functions will be assessed in different positions with the Cosmed Pony Fx Digital Spirometer (11). Forced vital capacity (FVC), forced expiratory volume in one second (FEV1), the ratio of forced expiratory volume in one second to forced vital capacity (FEV1/FVC), and peak expiratory flow rate (PEF) will be determined during the pulmonary function test.
Diagnostic Test: Fonseca Anamnestic Index — The questionnaire consists of 10 questions covering headaches, neck pain, temporomandibular joint pain, pain during chewing, parafunctional habits, malocclusion, and stress, and is scored as 10 (yes), 5 (sometimes), and 0 (no). The total score ranges from 0 to 100. A higher total score indicates an increased risk of temporomandibular joint problems.
Other: Jenkins Sleep Scale — The Jennkis Sleep Scale consists of four questions that assess sleep problems over a 4-week period. Each question is scored from 0 to 5. The total score ranges from 0 to 20 and indicates increasing sleep disturbance.
Other: Berlin Questionnaire — Berlin Questionnaire: The Berlin Questionnaire is a three-part assessment tool that assesses individuals' predisposition to sleep apnea. The first part contains five questions investigating snoring, the second part contains four questions investigating daytime sleepiness, and the third part contains two questions investigating hypertension and obesity. Each section is evaluated independently. Individuals who score 2 or higher in the first and second sections, and those who score 1 in the third section, are considered predisposed to sleep apnea. If two or more categories are positive, the participant is considered high risk for obstructive sleep apnea. If the participant scores two or more in the first and second categories, they are considered high risk. If blood pressure is high or BMI is above 30 kg/m2, the participant is considered high risk.
Other: Headache Impact Test-6 — Headache Impact Test-6: The Headache Impact Test-6 (HIT-6) is administered to identify activities individuals are unable to perform due to headaches and to determine the extent to which headaches impact daily life. This six-question questionnaire includes columns with increasing scores, from "never" to "always." Participants are asked to mark the box closest to their response. A high total score indicates that headaches negatively impact daily life.

SUMMARY:
The aim of the study was to evaluate the respiratory functions, sleep quality and headache severity of individuals with bruxism and to compare them with the control group without bruxism.

DETAILED DESCRIPTION:
Bruxism is defined as a repetitive jaw muscle activity characterized by teeth grinding or clenching accompanied by tooth wear and jaw muscle discomfort in the absence of a medical condition. Bruxism can occur during the day or during sleep and is defined as awake bruxism or sleep bruxism, respectively. According to the diagnostic criteria of the American Sleep Disorders Association (AASM), the New Classification of Sleep Disorders (ICSD-3), sleep bruxism requires the presence of a regular or frequent teeth grinding sound during sleep, accompanied by at least one of the following symptoms: signs of tooth wear, morning jaw fatigue or pain, and/or temporal headache and/or jaw locking. The etiology of bruxism is not fully understood but is influenced by psychosocial factors such as personality traits and stress. Sleep bruxism has been defined as a sleep-related movement disorder and has been reported to be associated with other sleep disorders. One sleep disorder reported to accompany bruxism is obstructive sleep apnea syndrome. Obstructive sleep apnea syndrome (OSAS) is characterized by upper airway obstruction that disrupts normal sleep patterns and ventilation despite respiratory efforts. OSAS is considered a risk factor for triggering bruxism. It has been suggested that rhythmic masticatory muscle activity during sleep bruxism plays a role in lubricating the upper gastrointestinal tract and increasing airway patency. This is assumed to facilitate better breathing. The possible relationship between sleep bruxism and sleep apnea suggests that the respiratory functions of individuals with bruxism may differ from those of individuals without bruxism. This difference is anticipated to be particularly pronounced in the supine sleep position. A review of the literature revealed no studies evaluating the respiratory functions of individuals with sleep bruxism. The study will also investigate sleep quality and headache severity in individuals with bruxism.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-45 years old

Exclusion Criteria:

* Receiving orthodontic or splint treatment

  * Having more than two missing teeth
  * Having undergone jaw, thoracic, or abdominal surgery within the last 6 months
  * Having a history of cervical and/or thoracic trauma
  * Having a neurological, systemic, and/or cardiopulmonary disease
  * Using sleeping pills
  * Having a diagnosis of psychiatric illness

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Male and female individuals between the ages of 18-45
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | From enrollment to the end of the assessment period at 2 hours
  Participant's forced vital capacity (FVC) will be assessed in different positions with the Cosmed Pony Fx Digital Spirometer. Forced vital capacity (FVC) is a subparameter of pulmonary function tests.
Forced expiratory volume in one second (FEV1) | From enrollment to the end of the assessment period at 2 hours
  Participants' forced expiratory volume in one second (FEV1) will be assessed in different positions with the Cosmed Pony Fx Digital Spirometer. Forced forced expiratory volume in one second (FEV1) is a subparameter of pulmonary function tests.
Peak expiratory flow rate (PEF) | From enrollment to the end of the assessment period at 2 hours
  Peak expiratory flow rate (PEF) will be assessed in different positions with the Cosmed Pony Fx Digital Spirometer. Peak expiratory flow rate (PEF) a subparameter of pulmonary function tests.

CONTACTS AND LOCATIONS:
Overall Officials: Seval Yılmaz, PhD., Principal Investigator — Atılım University
Locations (1):
- Atılım University, Ankara, Gölbaşı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share the data and it is collected for internal use only